CLINICAL TRIAL: NCT01596036
Title: Stages of Change Through the Cardiac Rehabilitation Experience After a Recent Hospitalization
Brief Title: Readiness for Behavior Change After a Heart Attack
Acronym: ENROLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Quinn R Pack, Cardiology Fellow, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HFHS 6649
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Myocardial Infarction; Stable Angina; Coronary Artery Disease
Keywords: cardiac rehabilitation; referral; enrollment; timing
MeSH Terms: conditions — Myocardial Infarction; Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Appointment (Experimental): Patients will receive an early appointment (within 10 days) from the time of their anticipated hospital discharge
  Interventions: Behavioral: Early appointment (within 10 days)
- Standard Referral (Placebo Comparator): Patients will receive an appointment to cardiac rehabilitation at 5 weeks from the date of their anticipated hospital discharge. A routine referral to cardiac rehabilitation will also occur in parallel. Consequently, it is possible that some patients will attend cardiac rehabilitation earlier than their assigned 5 week appointment.
  Interventions: Other: Routine referral (at 5 weeks)

INTERVENTIONS:
Behavioral: Early appointment (within 10 days) — Patients will receive an appointment to cardiac rehabilitation within 10 days from anticipated hospital discharge.
  Arms: Early Appointment
Other: Routine referral (at 5 weeks) — Standard Referral to Cardiac Rehabilitation
  Arms: Standard Referral

SUMMARY:
The purpose of this study is to test if an early appointment (within 10 days) when compared to a standard appointment (5 weeks) will affect attendance at the Cardiac Rehabilitation orientation and subsequent enrollment into cardiac rehabilitation.

DETAILED DESCRIPTION:
Cardiac Rehabilitation is central to full recovery after a myocardial infarction or a cardiac stenting procedure. Yet, this therapy is underutilized across the nation. Henry Ford currently enrolls about 42% of eligible patients. In addition, it currently takes, on average, 42 +/-26 days from hospital discharge to enrollment in rehabilitation. During this delay, there is strong tendency to return to prior habits (sedentary lifestyle, smoking, poor nutrition, etc.) that led to the myocardial infarction in the first place. This delay is both 1) unnecessary and 2) probably harmful to the patients' readiness to make changes.

The investigators seek to perform a randomized controlled trial of early (7-10 days) vs standard referral (5-6 weeks) to cardiac rehabilitation. In addition, the investigators will examine the patients' readiness to change through the first 3 months of the post-hospitalization period and correlate that to their behavior and enrollment in cardiac rehabilitation. Assessment of readiness to change will be accomplished by serial survey's, which will be administered at discharge, 2 weeks, 5 weeks, and 13 weeks after discharge.

Patients will consent to take the survey and be observed in a clinical study. However, in order to avoid the Hawthorne Effect, patients they will not initially be aware of the primary hypothesis, as the investigators strongly believe this will affect the main behavior they are trying to measure. Full patient disclosure will occur at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Stable Angina
* Myocardial infarction
* Percutaneous coronary intervention
* willingness to participate and consent for medical record review
* willingness to complete survey's

Exclusion Criteria:

* Recent illicit drug use
* Unstable psychiatric condition
* Moderate or severe dementia
* Inability to follow-up
* Leaving system with plans to enroll in cardiac rehabilitation out-of-system
* Inability to exercise (amputee, severe claudication)
* Unstable medical condition that would prevent regular exercise training
* Uncorrected severe aortic stenosis or severe mitral stenosis
* Referring physician feels that exercise is contra-indicated due to safety or other patient specific factors
* CABG, LVAD, or Heart Transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Attendance at the free orientation session for Cardiac Rehabilitation | within 5 weeks of randomized apointment date

SECONDARY OUTCOMES:
Completion of at least one exercise session in Cardiac Rehabilitation | within 1 month of orientation date
Total number of cardiac rehabilitation exercise sessions attended | within 6 months of actual orientation date
Completion of the cardiac rehabilitation program | within 6 months
  Completion is defined at attending the number of sessions agreed to at the onset of cardiac rehabilitation (e.g. agreeing to 3 session and attending 3) or attending 12 or more sessions.
Change in exercise capacity from the beginning to end of cardiac rehabilitation | within 6 months
  exercise capacity will be calculated from treadmill workloads using standardized formulas published in the 8th edition of ACSM's Guidelines for exercise testing and prescription
Readiness to make positive behavior changes | within 3 months
  Based on a 10 question survey, each patient will have a summary score to collapse across these questions. This summary score will be compared at 0, 5, and 13 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Quinn R Pack, MD, Principal Investigator — Henry Ford Hospital; Steven J Keteyian, PhD, Study Director — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

REFERENCES:
- [Background] Balady GJ, Ades PA, Bittner VA, Franklin BA, Gordon NF, Thomas RJ, Tomaselli GF, Yancy CW; American Heart Association Science Advisory and Coordinating Committee. Referral, enrollment, and delivery of cardiac rehabilitation/secondary prevention programs at clinical centers and beyond: a presidential advisory from the American Heart Association. Circulation. 2011 Dec 20;124(25):2951-60. doi: 10.1161/CIR.0b013e31823b21e2. Epub 2011 Nov 14. No abstract available. PMID 22082676
- [Background] Russell KL, Holloway TM, Brum M, Caruso V, Chessex C, Grace SL. Cardiac rehabilitation wait times: effect on enrollment. J Cardiopulm Rehabil Prev. 2011 Nov-Dec;31(6):373-7. doi: 10.1097/HCR.0b013e318228a32f. PMID 21826016
- [Derived] Pack QR, Mansour M, Barboza JS, Hibner BA, Mahan MG, Ehrman JK, Vanzant MA, Schairer JR, Keteyian SJ. An early appointment to outpatient cardiac rehabilitation at hospital discharge improves attendance at orientation: a randomized, single-blind, controlled trial. Circulation. 2013 Jan 22;127(3):349-55. doi: 10.1161/CIRCULATIONAHA.112.121996. Epub 2012 Dec 18. PMID 23250992